CLINICAL TRIAL: NCT01166880
Title: Imaging of Neonate Cerebral Vasculature
Brief Title: A Pilot Study Using Laser Speckle Imaging of Neonate Cerebral Vasculature
Status: Withdrawn | Type: Observational
Why Stopped: Unable to find grant fundingsupport to continue builds the study device.
Sponsor: University of California, Irvine (Other)
Collaborators: Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bernard Choi, Ph.D., Assistant Professor Biomedical Engineering, University of California, Irvine
Other Study IDs: 20097050
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Newborn Distress
Keywords: assessment
MeSH Terms: interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laser Speckle Imaging: Laser Speckle Imaging Infant Head Blood flow
  Interventions: Device: Laser Speckle Imaging

INTERVENTIONS:
Device: Laser Speckle Imaging — Laser Speckle Imaging Infant Head Blood flow

SUMMARY:
The researcher want to know whether reflections of light can be used to provide real-time pictures of blood vessel formation around infants' heads. This approach is called laser speckle imaging

DETAILED DESCRIPTION:
This study involves imaging of superficial blood vessels in the infant's head. Analysis of reflected light images provides the type of data necessary to see the blood vessels.

The researcher want to assess only feasibility of our instrument. If we determine that our instrument has sufficient spatial resolution to image directly large vessels, then we will proceed with plans for a larger study with statistical power.

ELIGIBILITY:
Inclusion Criteria:

* newborn

Exclusion Criteria:

* non-new bron

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: new born
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Neonate Cerebral Blood Flow | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Choi, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine